CLINICAL TRIAL: NCT03841812
Title: Comparation Analgesia Efficiency With Propofol Combine Sevoflurane vs Propofol Using Index of Nociception (NOX)
Brief Title: Comparation Analgesia Efficiency With Propofol Combine Sevoflurane vs Propofol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CINI-ZYLX-201809-50
Record Dates: First submitted 2019-01-19; First posted 2019-02-15 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-01

CONDITIONS: Nociceptive Pain; Analgesic Adverse Reaction; Inhalant Use
MeSH Terms: conditions — Nociceptive Pain | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Experimental): 5mg/kg/h Propofol continue infusion during the maintain of anesthesia during the maintain of anesthesia.
  Interventions: Drug: 5mg/kg/h Propofol
- Propofol & Sevoflurane (Experimental): 2mg/kg/h Propofol & 1% Sevoflurane group continue infusion(Balance anesthesia) during the maintain of anesthesia
  Interventions: Drug: Sevoflurane; Drug: 2 mg/kg/h Propofol

INTERVENTIONS:
Drug: 5mg/kg/h Propofol — 5mg/kg/h Propofol continuously infused during intre-operation
  Other Names: 5mg/kg/h Propofol Injection
  Arms: Propofol
Drug: Sevoflurane — 1% Sevoflurane continuously using during intre-operation.
  Other Names: 1% Sevoflurane
  Arms: Propofol & Sevoflurane
Drug: 2 mg/kg/h Propofol — 2mg/kg/h Propofol continuously infused during intre-operation
  Arms: Propofol & Sevoflurane

SUMMARY:
This study purpose to compare analgesia efficiency of propofol combine with sevoflurane with propofol only using index of Nociception (NOX)

DETAILED DESCRIPTION:
1. Recently study found sevoflurane plays an important role through spinal nerve peptide receptor (NK.1R), glycine receptor (GlyR), neuron nicotinic receptor (nnAChRs), Methyl-1-methyl-1-day aspartate (NMDA receptor), and TRPV1 receptor (TRPV1 receptor) produce the analgesic efficiency.
2. propofol was traditional sedation reagent.
3. index of Nociception (NOX) was the objective index for analgesia This study purpose to compare analgesia efficiency of Only Propofol and sevoflurane combine with propofol using index of Nociception (NOX)

ELIGIBILITY:
Inclusion Criteria:

* Participants were aged 18-65 years old,
* American Society of Anesthesiologists (ASA) physical status I, II or III
* scheduled to have urological surgery(would last longer than 1 h)
* requiring general anesthesia.

Exclusion criteria:

* refused to participate in this study;
* Unable to communicate normally because of consciousness alterations;
* a history of allergy to opioids
* contraindications to inhalational anesthesia
* a family history of malignant hyperthermia
* a history of alcohol or drug abuse
* received central nervous system-active drugs
* super obese as defined by a body mass index ≥40 kg/m2
* conditions liable to alter the pharmacokinetic and pharmacodynamic behaviors of the intravenous and inhalation anesthetics
* previous head injury
* neurologic
* psychiatric disease
* any disabling central nervous
* cerebrovascular disease
* using psychoactive
* anti-convulsive medications at the time
* unstable angina
* manifested congestive heart failure
* expected difficulty airway management

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
qNOX change | during operation
  Nociception of index (qNOX) difference between two groups. The nociception index (NOX) derived from electroencephalogram (EEG) signals has been proposed as a noninvasive guide to indicate anesthesia depth. The neurological processing of noxious stimuli is defined as nociception. NOX ranges from 0-99, and the lower the index, the deeper the state of analgesia. NOX lower than 20 represents deep analgesia, and higher than 80 represents inadequate analgesia.

SECONDARY OUTCOMES:
PACU duration | 24 hours
  Post anesthesia care unit duration(PACU duration). The longer PACU duration indicate the worse situation of the patients
PONV difference between two groups | 24 hours
  postoperative nausea and vomiting ratio(PONV) difference between two groups. The more frequency of PONV, the worst comfortable outcome of the patients
Post- operative pain difference between two groups | 24 hours
  Post- operative pain difference between two groups using VAS(Visual analogue rating) Score evaluation. Pain was assessed 24 h post operation using a 0-10 numeric pain rating scale (VAS scale), where zero meant no pain and 10 meant the worst imaginable pain.VAS score (Post-operation 24 h) (0-1 VAS indicate None pain; 2-5 VAS indicate Moderate pain; 6-10 VAS indicate severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Ke Huang, MS, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China